CLINICAL TRIAL: NCT04664192
Title: Bio-Banking of Specimens for Advanced Lung Disease and Lung Transplant Research
Acronym: ALD Biobank
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Susan Mathai, Pulmonary Disease specialist, Baylor Research Institute
Other Study IDs: 021-007
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Failure; Interstitial Lung Disease; Lung Diseases
MeSH Terms: conditions — Respiratory Insufficiency; Lung Diseases, Interstitial; Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, serum samples, plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung transplant Recipients: Biobank registry for Lung transplant recipients
  Interventions: Other: Patient Biospecimen Registry (observational and blood sampling)

INTERVENTIONS:
Other: Patient Biospecimen Registry (observational and blood sampling) — Clinical data collected at every blood sample collection visit.

SUMMARY:
A major goal of this protocol is to support biomarker studies in advanced lung diseases, lung transplantation care, and to improve our understanding of the effects of viral and other infectious exposures to outcomes in our lung transplant and ALD patient populations.

DETAILED DESCRIPTION:
The identification of biomarkers in a patient's blood or tissue that are specific for particular medical conditions (such as interstitial lung disease, chronic obstructive lung disease (COPD), and post-lung transplant rejection) is important for the prevention and early detection of the disease, as well as to advance our understanding of targeted therapies. Availability of biomarkers for diagnosis and for the prediction of patient prognosis and therapy promises personalized medicine. Patients may be selected based on the presence of particular gene mutations or circulating protein levels to receive personalized treatment. Furthermore, knowledge regarding genetic risk and susceptibility to infectious diseases as well as structural lung disease is rapidly growing-as whole genome sequencing and genome-wide association studies have become easier to do, genetic risk has emerged as increasingly important in understanding why and how some patients develop chronic lung disease. This is true for the spectrum of lung diseases treated in the ALD program, from those with airways diseases such as COPD to diffuse parenchymal lung diseases such as idiopathic pulmonary fibrosis (IPF). The availability of human biological specimens for research purposes is crucial for the advancement of medical knowledge of understanding, diagnosing, and treating chronic lung diseases and optimizing post-lung transplant care.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals aged 18 years and older
2. Persons who have undergone lung transplantation at Baylor University Medical Center in the previous 10 years
3. Individual is able to understand and sign the informed consent form

Exclusion Criteria:

1. Significant documented anemia (hemoglobin <8 g/dL)
2. Blood transfusions within past 3 weeks
3. Active cancer (non-skin cancers)
4. Enrollment against doctor recommendation
5. Patient not able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of patients with lung transplant | 5 years
  ICD 10 code for underlying lung disease

SECONDARY OUTCOMES:
Survival | 5 years
  Date of death

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mathai, MD, Principal Investigator — Baylor Scott & White Research Institute
Locations (1):
- Baylor Scott & White Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No